CLINICAL TRIAL: NCT02833688
Title: the Ethnic Committee of the Chinese People's Liberation Army (PLA) General Hospital
Brief Title: Effects of Dexmedetomidine on the Liver Injury After Hepatectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yu Zhang, attending doctor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PLAGHAOC00***
Record Dates: First submitted 2016-07-05; First posted 2016-07-14 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Ischemia-reperfusion Injury
MeSH Terms: conditions — Reperfusion Injury | interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dexmedetomidine (Experimental): dexmedetomidine 2mg is diluted in 0.9% sodium chloride with the concentration of 4 ug ml-1 is administered with an loading dose of 0.5ug kg-1 of 10 min, and maintained with infusion rate of 0.5 ug kg-1 h-1. The infusion is ceased after the resection of the hepatic issues.
  Interventions: Drug: dexmedetomidine
- 0.9% sodium chloride (Placebo Comparator): 0.9% sodium chloride is administered with an loading dose of 0.5ug kg-1 of 10 min, and maintained with infusion rate of 0.5 ug kg-1 h-1. The infusion is ceased after the resection of the hepatic issues.
  Interventions: Drug: 0.9% sodium chloride

INTERVENTIONS:
Drug: dexmedetomidine — dexmedetomidine 2mg is diluted in 0.9% sodium chloride with the concentration of 4 ug ml-1 is administered with an loading dose of 0.5ug kg-1 of 10 min, and maintained with infusion rate of 0.5 ug kg-1 h-1. The infusion is ceased after the resection of the hepatic issues.
  Arms: dexmedetomidine
Drug: 0.9% sodium chloride — 0.9% sodium chloride is administered with an loading dose of 0.5ug kg-1 of 10 min, and maintained with infusion rate of 0.5 ug kg-1 h-1. The infusion is ceased after the resection of the hepatic issues.
  Arms: 0.9% sodium chloride

SUMMARY:
To investigate whether dexmedetomidine reduce liver injury after hepatectomy. During hepatectomy, surgeons always took inflow occlusion to reduce blood loss with Pringle maneuver. A few clinical studies had shown dexmedetomidine could reduce ischaemia/reperfusion (IR) injury caused by the secretion of reactive oxygen species and inflammatory cytokines. Glutathione-S-transferase (GST) was a sensitive and specific marker for hepatic injury in several studies before. So the investigator decided to use it as the primary endpoint. Besides, in our center, there are some liver resection surgeries that didn't need occlusion. So it can serve the best placebo for determine the the actual effect of dexmedetomidine on the IR injury in further subgroup analysis.

DETAILED DESCRIPTION:
The purpose of our study is to compare liver injury with dexmedetomidine. The enrolled patients were randomized into two group. In the study group, dexmedetomidine, diluted in 0.9% sodium chloride with the concentration of 4 ug ml-1 is administered with an loading dose of 0.5ug kg-1 of 10 min, and maintained with infusion rate of 0.5 ug kg-1 h-1. While, 0.9% sodium chloride serves as the placebo with the same loading dose and infusion rate in the control group. The infusion is ceased after the resection of the hepatic issues.

GST is a sensitive and specific marker for hepatic injury in several studies before and is taken as the primary endpoint. And the investigator use other inflammatory cytokines reflecting the systemic inflammatory response in serum. Besides these, the investigator observe the hemodynamic changes during the operation time and complications related with anesthesia and surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) I~III
* selected to have hepatectomy in our hospital, Child-Pugh A
* patient's consent

Exclusion Criteria:

* refusing to attend or attending in other clinical study
* having severe cardio-pulmonary disease, ejection fraction (EF)<40%, having cardiac infarction in recent three months, chronic obstructive pulmonary disease (COPD) (PaO2<60mmHg)
* pregnant or lactating women
* having neuropsychiatric disorders
* emergent surgeries，hemorrhage shock，
* rupture and hemorrhage of liver tumor

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-08-02 (Actual); Primary Completion 2017-01-26 (Actual); Study Completion 2017-01-26 (Actual)

PRIMARY OUTCOMES:
GST | 24 hours
  baseline (before the surgery), 30 minutes after hepatic resection, 1 day after hepatectomy 30 minutes after hepatic resection

SECONDARY OUTCOMES:
interleukin (IL-6), tumor necrosis factor (TNF-a) | 24 hours
  baseline (before the surgery), 30 minutes after hepatic resection, 1 day after hepatectomy

OTHER OUTCOMES:
Complications after surgery | 1 month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Weidong MI, Doctor, Study Chair — CHINA
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided